CLINICAL TRIAL: NCT04276857
Title: Systemic Therapy With a Loco-regional Treatment in Patients With Locally Advanced Pancreatic Cancer: The SMART Study
Brief Title: Systemic Therapy With a Loco-regional Treatment in Patients With Locally Advanced Pancreatic Cancer
Acronym: SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Shahid Ahmed, Professor of Medicine, University of Saskatchewan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 284
Record Dates: First submitted 2019-11-08; First posted 2020-02-19 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Locally Advanced Pancreatic Cancer; Irreversible Electroporation
MeSH Terms: interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm study (Other): All eligible patients will receive combination chemotherapy and if there i s a positive response they will undergo IRE.
  Interventions: Device: Irreversible electroporation (NanoKnife® )

INTERVENTIONS:
Device: Irreversible electroporation (NanoKnife® ) — IRE is a unique treatment modality as it ablates tumor cells without using heat or radiation and hence does not cause injury to nearby blood vessels, ducts, and bowel. This makes it particularly appealing for the treatment of locally advanced unresectable pancreatic cancers. This local treatment for cancer involves delivering brief pulses of high voltage electrical current across the tumor (either percutaneously or open surgery), which results in the formation of tiny holes (nanopores) in the cell membranes.
  Other Names: FOLFIRINOX (5-FU, leucovorin, irinotecan, and oxaliplatin) or gemcitabine/nab-paclitaxel

SUMMARY:
Background

Pancreatic cancer is one the leading causes of cancer-related death in Canada. Approximately 40 percent of patients with pancreatic cancer present with locally advanced pancreatic cancer and are not candidate for curative surgery. The optimal management of patients with locally advanced pancreatic cancer remains unknown. Most patients are treated with chemotherapy alone and role of local treatment such as radiation is not well defined. Other conventional ablative therapies such as thermal ablation and cryoablation have limited role in locally advanced pancreatic cancer due to the risk of collateral damage to the adjacent structures. Irreversible electroporation (IRE) is a novel non-thermal ablation technology that does not cause injury to nearby blood vessels, ducts, and bowel and has potential to provide longer disease control and thereby a better overall survival. The current study aims to prospectively validate effectiveness and safety of IRE in real-world patients with locally advanced pancreatic cancer.

Objectives

1) To determine 12-month progression-free survival (PFS) and 24-month overall survival rates of patients with locally advanced pancreatic cancer who are treated with combination chemotherapy and IRE and 2) to compare progression-free and overall survival of patients with locally advanced pancreatic cancer who are treated with combination chemotherapy and IRE versus combination chemotherapy alone.

Design

Prospective multicenter single arm study.

Methods

Based on the assumption of doubling of PFS of patients who are being treated with IRE and chemotherapy versus chemotherapy alone we estimated a sample of n=27 of adult patients with histologically proven non-metastatic locally advanced adenocarcinomas. Eligible patients will be recruited at the two major cancer centers in Saskatchewan. All IRE eligible patients will receive 12 weeks of induction chemotherapy and will undergo repeat imaging studies. If there is no disease progression IRE will be performed. An additional 12 weeks of chemotherapy will be recommended. Patients who are not eligible for IRE due to size criteria will receive chemotherapy at the discretion of treating oncologist till disease progression or till they become eligible for IRE. Quality of life will be assessed every three months or until disease progression.

Significance

Despite progress in the management of most solid organ cancers and better outcomes, little advancement has been made in the treatment of patients with locally advanced pancreatic cancer. Unfortunately, most patients have very limited life expectancy. There is an unmet need for novel approaches in the management of patients with locally advanced pancreatic cancer. IRE in combination with chemotherapy has potential to improve local disease control and thereby improves survival and may prove a valuable tool to add in the multidisciplinary treatment of cancer. The result of this study will be used for the development of a future multicenter national phase III trials.

DETAILED DESCRIPTION:
Current Knowledge and Rationale

Pancreatic cancer is one of the most lethal malignancies, with an overall 5-year survival rate of less than 10%. It is the 12th most common cancer and 7th most frequent cause of cancer-related death worldwide and 4th leading cause of cancer death among men and women in Canada. Surgery is the only curative option, however, less than 20% of patients have resectable disease at the time of diagnosis and the remainder have either locally advanced or metastatic cancer. Approximately 40 percent of patients with pancreatic cancer present with locally advanced or surgically unresectable pancreatic cancer. The optimal management of patients with locally advanced pancreatic cancer remains unknown. Treatment options include chemotherapy alone, radiation alone, or combination of chemotherapy and radiation. Despites absence of metastatic disease at the time of diagnosis, patients with locally advanced pancreatic cancer have poor prognosis with a median overall survival of about 12 months.

For many years single agent gemcitabine remained the standard therapy for patients with locally advanced and metastatic pancreatic cancer (6). Two randomized trials showed benefit of combination chemotherapy over single agent gemcitabine. For example, the ACCORD II trial demonstrated the efficacy of FOLFIRINOX (5-FU, leucovorin, irinotecan, and oxaliplatin) over gemcitabine in patients with metastatic pancreatic cancer. The median progression-free survival (PFS) and overall survival (OS) with FOLFIRNOX were 6.4 months and 11.1 months, respectively, compared with 3.3 months and 6.8 months, respectively, with gemcitabine alone. The MPACT trial demonstrated the superiority of the combination of gemcitabine plus nab-paclitaxel over gemcitabine alone in patients with metastatic pancreatic cancer. The median PFS and OS were 5.5 months and 8.5 months, respectively, in the gemcitabine/nab-paclitaxel group, compared with 3.7 and 6.7 months in the gemcitabine group, respectively. Based on the improved activity and survival of both regimens in patients with metastatic pancreatic cancer, FOLFIRINOX (5-FU, leucovorin, irinotecan, and oxaliplatin) and gemcitabine plus nab-paclitaxel have become standard chemotherapy regimens in the management of patients with locally advanced pancreatic cancer. In the investigators' world experience of patients with locally advanced pancreatic cancer who were treated with either FOLFIRINOX (5-FU, leucovorin, irinotecan, and oxaliplatin) or gemcitabine plus nab-paclitaxel over a five year period in Saskatchewan had a median OS of 12.0 months.

Because patients with locally advanced pancreatic cancer have localized disease, loco-regional therapies such as radiation treatment have been employed with limited success. For example, in a randomized trial involving 449 patients with locally advanced pancreatic cancer with stable disease after 4 months of induction chemotherapy, there was no significant difference in overall survival with chemoradiotherapy compared with chemotherapy alone. The median OS of patients who received chemotherapy was 16.5 months compared with 15.2 months it combination of chemotherapy and radiation (p=0.83). Currently, in most institutions outside the setting of a clinical trial, patients with locally advanced pancreatic cancer, are primarily treated with combination of chemotherapy. Other conventional ablative therapies such thermal ablation have limited role due to collateral damage to the adjacent vital structure such as blood vessels and bile duct. These limitations could be overcome by irreversible electroporation (IRE), a novel, non-thermal ablative method that has been examined in the treatment of various solid organ cancers.

IRE also known as NanoKnife® is a unique treatment modality as it ablates tumor cells without using heat or radiation and hence does not cause injury to nearby blood vessels, ducts, and bowel. This makes it particularly appealing for the treatment of locally advanced unresectable pancreatic cancers. This local treatment for cancer involves delivering brief pulses of high voltage electrical current across the tumor (either percutaneously or open surgery), which results in the formation of tiny holes (nanopores) in the cell membranes. The loss of electrolytes and the gain of fluid into the cell from these pores causes the cells to die an apoptotic death. The collagen scaffolding is unaffected because IRE ablation occurs without heat, and this allows for destruction of tumors without collateral thermal injury. IRE is therefore an ideal ablation strategy for the pancreas, which is intimate with the common bile duct, the portal vein, and the duodenum, all of which are injured if heat ablation or even radiation are used.

IRE has been evaluated in patients with hepatobiliary and pancreatic tumors. Currently most results about efficacy and safety of IRE are derived from retrospectives studies and case series. The largest retrospective series about IRE involving 200 patients with locally advanced pancreatic cancer is reported by Martin and others. In their study the addition of IRE to conventional chemotherapy and radiation therapy resulted in prolonged survival compared with historical controls. With a median follow-up of 29 months, median OS of treated cohort was 24.9 months . Among them 37% experienced complications but most were mild to moderate. A recent retrospective study involving 50 patients with locally advanced pancreatic cancer is reported by Narayanan and others. Median OS of study cohort was 27.0 months from time of diagnosis and 14.2 months from time of IRE. Of note, patients with 3 cm or smaller tumors had better survival. There was no IRE-related mortality. Serious adverse events occurred in 20% patients. Despite promising results with IRE in patients with locally advanced pancreatic cancer, currently, there is a very limited prospective data available. The current study aims to prospectively validate efficacy and safety of IRE in Canadian patients with locally advanced pancreatic cancer and based on the result develop a later phase multicenter national clinical trial.

Primary Research question

Does addition of IRE to combination of chemotherapy in patient with locally advanced pancreatic cancer improve their outcomes?

Hypothesis

It is hypothesized that addition of IRE to combination of chemotherapy in patients with locally advanced pancreatic cancer improves median PFS from 4-6 months to 10-12 months and median OS from 12 months to approximately 24 months.

Methods

Study Design and Sample Size The SMART study is a prospective multicenter single arm phase II study. Assuming 12-month disease progression rate of 40% in patients treated with IRE and chemotherapy versus 80% in patients who are treated with chemotherapy alone a sample of n=27 to achieve 80% power with an alpha error of 0.05 is estimated. The eligible patients will be recruited over a two-year period at the two major cancer centers in Saskatchewan.

Assessment, interventions, and follow-up visits Potentially eligible patients will be identified by the provincial hepatobiliary surgical team and will be discussed in a multidisciplinary hepatobiliary-pancreatic cancer round. Patients with locally advanced pancreatic cancer will be assessed by a medical oncologist and if are found to be eligible for combination chemotherapy will be offered the study. Eligible patients will receive 3 months of FOLFIRINOX or Gemcitabine plus nab-paclitaxel at the discretion of treating oncologist (induction phase). Treatment will be administered in an out-patient chemotherapy unit. Baseline and follow up imaging studies will be performed as per current standard (CT scan every 2-3 months and PET and other imaging studies as indicated). The candidacy for the procedure will be determined by IRE team comprised of diagnostic radiologist, interventional radiologist, hepatobiliary surgeon and a medical oncologist. Patients who do not progress following induction chemotherapy and are candidate for IRE will undergo IRE.

Approximately four weeks after the procedure patients will be assessed by the treating oncologist and 3 additional months of chemotherapy will be recommended. After total six months of chemotherapy if there is no progression further chemotherapy could be given at the discretion of treating physicians. Those patients who are not found to be eligible for IRE will continue to receive chemotherapy (continuation phase). Their scans will be reviewed every 2-3 months by the IRE team for potential eligibility for IRE till disease progression. Quality of life will be assessed at baseline, after induction chemotherapy, and prior to the start of second phase of chemotherapy and then every three months till disease progression. Periodic assessment prior to each cycle of chemotherapy, blood work and imaging study will be performed as per standard for pancreatic cancer. Specific drug reductions and management of side effects will be in accordance with published recommendations and will be at the discretion of treating oncologists. On progression patients will be off the study. All patients will be followed at the cancer center till their death.

Analysis Response rates and stable disease rates will be summarized by percentages and their 95% CI. Survival curves will be analyzed using the Kaplan-Meier method, and differences between groups will be analyzed using log-rank test. The efficacy and toxicities of IRE will be recorded and be compared with the historic control from the publish literature. In addition, a subgroup of patients who are no able to undergo IRE will serve as an internal control. Correlation will be significant at the .05 level (two tailed). A Cox proportional survival analysis will be done to assess various clinical and pathologic factors for their correlation with survival.

Quality of Life:

The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) along with the EORTC Pancreatic Cancer Module (QLQ-PAN26). The EORTC QLQ-C30 is a widely used instrument for measuring general cancer QOL. It consists of 30 items and patients responses are transformed to produce 0-100 scores on five functional scales, nine symptom scales and a scale representing global quality of life. Higher functional scale scores indicate better QOL whereas higher symptom scale/item scores indicate higher level of symptoms. The QLQ-PAN26 is currently being validates for patients with pancreatic cancer. The QOL will be measured periodically as described above.

Correlative science

Five cc blood will be collected and freeze at baseline and after induction phase of chemotherapy, (0 and 3 months) and within 4 weeks and 12 weeks (0 and 3 months) after IRE for patients who undergo IRE for future correlative science study.

Timeline

Each year about 160 patients are diagnosed with pancreatic cancer in Saskatchewan. About 40% of them have locally advanced pancreatic cancer. Assuming 40% of patients with newly diagnosed locally advanced pancreatic cancer are eligible for combination chemotherapy (FOLFIRINOX or gemcitabine Nab paclitaxel), accrual was estimated at a rate of 1-2 patient per month over a period of 18-24 months. In Saskatchewan all patients with locally advanced pancreatic cancer are followed for indefinite period of time at the cancer center. After the two-year period patients who are on active treatment or in remission following IRE will continue to be follow for progression-free and overall survival.

Knowledge Translation

The research findings will be presented in the international cancer conferences and published in peered review journals. In addition, following strategies will be used to facilitate knowledge dissemination and its application.

* The results will be shared with the knowledge users using various platforms at the different stages of research (tumor-groups meetings/rounds, cancer conferences, guideline/clinical trials meetings, newsletter, etc.).
* The results will be presented to the Pharmacy and Therapeutic Committee of Saskatchewan for implementation of research findings.
* Networking and communication will be done with the Western and Eastern Canadian Gastrointestinal Cancer groups to share results and to work on developing a late phase clinical trial.

Significance

Despite progress in the management of most solid organ cancers and better outcomes, little advancement has been made in the treatment of patients with locally advanced pancreatic cancer. Unfortunately, most patients have very limited life expectancy. There is an unmet need for novel approaches in the management of patients with locally advanced pancreatic cancer. IRE in combination with chemotherapy has potential to improve local disease control and thereby improves survival previously and may prove a valuable tool to add in the multidisciplinary treatment of cancer. This approach in combination of chemotherapy could potentially be more cost effective than continuing chemotherapy alone. In addition, in the proposed study patients selection for their eligibility of combination chemotherapy and dose modification will be at the discretion of treating oncologists. This approach will broaden generalizability of the results and will provide a real-world experience. It is expected that the result of this study will guide for the development of a future multicenter national late phase trial.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with biopsy-proven locally advanced pancreatic adenocarcinoma who are candidates for combination chemotherapy as determined by treating oncologists.

Exclusion Criteria:

1. Pregnancy
2. Metastatic pancreatic cancer
3. Another active second primary cancer with the exception of squamous cell carcinoma of the skin or an in situ cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
1 year progression free survival rate of patients with locally advanced pancreatic cancer who are treated with IRE and combination chemotherapy. | At 12 months after enrollment into the study
  Progression free survival

SECONDARY OUTCOMES:
2 years overall survival rate of patients with locally advanced pancreatic cancer who are treated with IRE and combination chemotherapy. | At 2 years after enrollment into the study
  Overall survival
quality of life of patients with locally advanced pancreatic cancer who are treated with combination chemotherapy and IRE: EORTC QOL 30 | Every 3 months
  EORTC QOL 30, Raw scores are transformed to a 0-100 scale, with higher scores representing better functioning/QOL and greater symptom burden
12 and 24 months rate of IRE in patients with locally advanced pancreatic cancer who are initially deemed to be ineligible for IRE. | At 12 and 24 months
  IRE rate
30-day and 90-day complications rate of IRE. | 30 and 90 days
  Complication
cost-effectiveness of IRE in patients with locally advanced pancreatic cancer. | At 2 years
  Cost-effectiveness
compare progression-free and overall survival of sub-groups of patients with locally advanced pancreatic cancer who are treated with combination chemotherapy and IRE versus combination chemotherapy alone. | At 2 years
  PFS and overall survival
Prognostic significance of circulating DNA | At 3 years
  correlation between circulating DNA and progression-free and overall survival of patients with locally advanced pancreatic cancer who are treated with combination IRE and or chemotherapy.
Prognostic bio-markers | At 3 years
  A panel of 47 genes using next generation sequencing technique

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Ahmed, MD, PhD, Principal Investigator — University of Saskatchewan
Locations (2):
- Canada (2):
  - Allan Blair Cancer Center, Regina, Saskatchewan
  - Saskatoon Cancer Center, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided
due to confidentiality it may not be feasible

REFERENCES:
- [Background] Hidalgo M. Pancreatic cancer. N Engl J Med. 2010 Apr 29;362(17):1605-17. doi: 10.1056/NEJMra0901557. No abstract available. PMID 20427809
- [Background] Vincent A, Herman J, Schulick R, Hruban RH, Goggins M. Pancreatic cancer. Lancet. 2011 Aug 13;378(9791):607-20. doi: 10.1016/S0140-6736(10)62307-0. Epub 2011 May 26. PMID 21620466
- [Background] International Cancer facts and figures. Pancreatic cancer statistics. http://www.wcrf.org/int/cancer-facts-figures/data-specific-cancers/pancreatic-cancer-statistics (accessed on July 10th 2017).
- [Background] Canadian Cancer Statistics 2016. http://www.cancer.ca/~/media/cancer.ca/CW/cancer%20information/cancer%20101/Canadian%20cancer%20statistics/Canadian-Cancer-Statistics-2016-EN.pdf?la=en (Accessed on July 13th, 2017).
- [Background] Balaban EP, Mangu PB, Khorana AA, Shah MA, Mukherjee S, Crane CH, Javle MM, Eads JR, Allen P, Ko AH, Engebretson A, Herman JM, Strickler JH, Benson AB 3rd, Urba S, Yee NS. Locally Advanced, Unresectable Pancreatic Cancer: American Society of Clinical Oncology Clinical Practice Guideline. J Clin Oncol. 2016 Aug 1;34(22):2654-68. doi: 10.1200/JCO.2016.67.5561. Epub 2016 May 31. PMID 27247216
- [Background] Burris HA 3rd, Moore MJ, Andersen J, Green MR, Rothenberg ML, Modiano MR, Cripps MC, Portenoy RK, Storniolo AM, Tarassoff P, Nelson R, Dorr FA, Stephens CD, Von Hoff DD. Improvements in survival and clinical benefit with gemcitabine as first-line therapy for patients with advanced pancreas cancer: a randomized trial. J Clin Oncol. 1997 Jun;15(6):2403-13. doi: 10.1200/JCO.1997.15.6.2403. PMID 9196156
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Papneja N, Zaidi A, Chalchal H, Moser M, Tan K, Olson C, Haider K, Shaw J, Ahmed S. Comparisons of Outcomes of Real-World Patients With Advanced Pancreatic Cancer Treated With FOLFIRINOX Versus Gemcitabine and Nab-Paclitaxel: A Population-Based Cohort Study. Pancreas. 2019 Aug;48(7):920-926. doi: 10.1097/MPA.0000000000001340. PMID 31180981
- [Background] Hammel P, Huguet F, van Laethem JL, Goldstein D, Glimelius B, Artru P, Borbath I, Bouche O, Shannon J, Andre T, Mineur L, Chibaudel B, Bonnetain F, Louvet C; LAP07 Trial Group. Effect of Chemoradiotherapy vs Chemotherapy on Survival in Patients With Locally Advanced Pancreatic Cancer Controlled After 4 Months of Gemcitabine With or Without Erlotinib: The LAP07 Randomized Clinical Trial. JAMA. 2016 May 3;315(17):1844-53. doi: 10.1001/jama.2016.4324. PMID 27139057
- [Background] Deipolyi AR, Golberg A, Yarmush ML, Arellano RS, Oklu R. Irreversible electroporation: evolution of a laboratory technique in interventional oncology. Diagn Interv Radiol. 2014 Mar-Apr;20(2):147-54. doi: 10.5152/dir.2013.13304. PMID 24412820
- [Background] Ruarus AH, Vroomen LGPH, Puijk RS, Scheffer HJ, Zonderhuis BM, Kazemier G, van den Tol MP, Berger FH, Meijerink MR. Irreversible Electroporation in Hepatopancreaticobiliary Tumours. Can Assoc Radiol J. 2018 Feb;69(1):38-50. doi: 10.1016/j.carj.2017.10.005. PMID 29458954
- [Background] Scheffer HJ, Nielsen K, de Jong MC, van Tilborg AA, Vieveen JM, Bouwman AR, Meijer S, van Kuijk C, van den Tol PM, Meijerink MR. Irreversible electroporation for nonthermal tumor ablation in the clinical setting: a systematic review of safety and efficacy. J Vasc Interv Radiol. 2014 Jul;25(7):997-1011; quiz 1011. doi: 10.1016/j.jvir.2014.01.028. Epub 2014 Mar 18. PMID 24656178
- [Background] Al Efishat M, Wolfgang CL, Weiss MJ. Stage III pancreatic cancer and the role of irreversible electroporation. BMJ. 2015 Mar 18;350:h521. doi: 10.1136/bmj.h521. PMID 25787829
- [Background] Martin RC 2nd, Kwon D, Chalikonda S, Sellers M, Kotz E, Scoggins C, McMasters KM, Watkins K. Treatment of 200 locally advanced (stage III) pancreatic adenocarcinoma patients with irreversible electroporation: safety and efficacy. Ann Surg. 2015 Sep;262(3):486-94; discussion 492-4. doi: 10.1097/SLA.0000000000001441. PMID 26258317
- [Background] Narayanan G, Hosein PJ, Beulaygue IC, Froud T, Scheffer HJ, Venkat SR, Echenique AM, Hevert EC, Livingstone AS, Rocha-Lima CM, Merchan JR, Levi JU, Yrizarry JM, Lencioni R. Percutaneous Image-Guided Irreversible Electroporation for the Treatment of Unresectable, Locally Advanced Pancreatic Adenocarcinoma. J Vasc Interv Radiol. 2017 Mar;28(3):342-348. doi: 10.1016/j.jvir.2016.10.023. Epub 2016 Dec 16. PMID 27993507